CLINICAL TRIAL: NCT01497977
Title: Impact of Phytoestrogens on Serum Lipids in Postmenopausal Women
Brief Title: Phytoestrogen Supplementation in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Medical Academy, Serbia (Other)
Responsible Party: Principal Investigator, Tihomir Mihailovic, Dr, American Medical Academy, Serbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 175062
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Low Serum Lipid Levels
Keywords: phytoestrogens; postmenopause; serum lipids
MeSH Terms: interventions — Phytoestrogens; Isoflavones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- soya phytoestrogens (Experimental)
  Interventions: Drug: phytoestrogens
- red clover phytoestrogens (Experimental)
  Interventions: Drug: phytoestrogens
- No drugs (No Intervention)

INTERVENTIONS:
Drug: phytoestrogens — The red clover capsule consisted of 4 isoflavones: biokain A (23mg), daidzein (1mg), formononetin (15mg) and genistein (1mg).
  Other Names: isoflavones
  Arms: red clover phytoestrogens
Drug: phytoestrogens — The soya daily dose contained 2 isoflavones: genistein (39mg) and daidzein (1mg).
  Other Names: isoflavones
  Arms: soya phytoestrogens

SUMMARY:
The goal of the study was to assess the impact of soy and red clover derived phytoestrogens on serum lipids in postmenopausal women. Both soya and red clover have high phytoestrogen content. Phytoestrogens, a class of estrogenic molecules produced by plants bind to the estrogen receptor and are capable of producing estrogenic effects. Therefore, our hypothesis was that they can reduce the levels of serum lipids.

Materials and Methods: Researchers investigated total cholesterol, cholesterol fractions and triglycerides in blood, before treatment and in six months periods, throughout 18 months. The study involved 74 healthy postmenopausal women, divided into three groups. The first group of 23 patients received red clover derived isoflavones, the second one with 26 patients got soy derived phytoestrogens, while the third, control group with 25 patients, was without medications.

DETAILED DESCRIPTION:
A classic clinical sample was constructed. A total of 117 consecutive postmenopausal women who came to us in four months periods due to the postmenopausal symptoms (hot flushes, sleep disturbances, mood swings and vaginal dryness) were enlisted for the research. Out of them 74 fulfilled the inclusion criteria and were randomized. Randomization process was simple manual and was done in the way that every woman with the odd randomization number received soya while those with the even randomization number received red clover derived isoflavones. However, during the study neither the doctors nor the patients knew what the randomization was and what the medication was. Women in the control group did not receive any medications and were only used for comparison. Examinees for this group were randomly selected from healthy postmenopausal women who had regular colposcopic check-ups during the same period. Out of 186 such women, 111 fulfilled the inclusion criteria, and every third was recruited for the study. In such way patients have been randomly divided in three groups (soya - S, red clover - RC, control - C) consisting of 37 women each. However, 6 women had to be excluded from soya and 5 from red clover group, as they did not take treatment on regular basis. Moreover, 7 women from soya, 6 from red clover and 9 from control group were excluded as a result of developing health problems (hypertension in 11 cases and uterine bleeding in 8 cases and H-SIL in 3 cases). One woman from soya group wanted to start taking hormone replacement therapy. Three women decided to drop out from the control group. So, finally 23 women from soya group, 26 from red clover and 25 from control group had undergone the study to the end.

Women were taking one capsule per day of either soya or red clover derived phytoestrogens, early in the morning, before meal. The soya daily dose contained 2 isoflavones: genistein (39mg) and daidzein (1mg), while the red clover capsule consisted of 4 isoflavones: biokain A (23mg), daidzein (1mg), formononetin (15mg) and genistein (1mg). Each patient was keeping self-reported daily diary of the therapy administration, symptoms and adverse reactions.

Researchers investigated total cholesterol, cholesterol fractions (LDL, HDL) and triglycerides, in cubital vein blood of patients, as well as body height and weight for each subject (out of which Body Mass Index - BMI was calculated by the standard formula). Data were recorded at the study beginning and 6, 12 and 18 months after the treatment commencement. Standard tests for lipid level evaluation were carried out on Olympus AU 400 automatic analyzer with referral rates for triglycerides from 0,61 to 2,10 mmol/l, total cholesterol 3,63 - 6,46 mmol/l, HDL 0,75 - 1,99 mmol/l, LDL 1,60 - 4,78 mmol/l.

ELIGIBILITY:
Inclusion Criteria:

* healthy postmenopausal women, not taking any medications (anti-osteoporotic, lipid-lowering, anti-hypertensive and hormone based) that could influence the study results, last menstrual cycle of the investigated women was at least 12 months before entering the study.

Exclusion Criteria:

* unfulfilled inclusion criteria at any time of the study, allergies or severe adverse reactions on the administered drugs, changing of the regular dietary habits, the study protocol interruption and the wish of the patient to withdraw from the study.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline of serum lipids | 18 months
  study begining, 6 months, 12 months, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Tihomir Mihailovic, MD.PhD, Study Director — Ultramedica Clinic, American Medical Academy; Milan Terzic, Prof. dr, Principal Investigator — School of Medicine, University of Belgrade
Locations (1):
- Ultramedica Clinic, American Medical Academy, Belgrade, Serbia